CLINICAL TRIAL: NCT03370991
Title: Blueberry Consumption for Improving Vascular Endothelial Dysfunction in Postmenopausal Women With Elevated Blood Pressure and Stage 1-Hypertension
Brief Title: Blueberries for Improving Vascular Endothelial Function in Postmenopausal Women With Elevated Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Principal Investigator, Sarah Johnson, Assistant Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1255927
Record Dates: First submitted 2017-12-02; First posted 2017-12-13 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Menopause; Elevated Blood Pressure; Hypertension; Endothelial Dysfunction
Keywords: Blueberries; Polyphenols; Cardiovascular Disease; Atherosclerosis; Oxidative Stress; Inflammmation; Endothelium; Vasodilation; Blood Pressure; Menopause; Women's Health; Functional Food; Bioactive Compounds; Dietary Supplements; Aging
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Atherosclerosis; Aneurysm

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry (Experimental): 22 g/day freeze-dried blueberry powder for 12 weeks
  Interventions: Dietary Supplement: Blueberry Powder
- Control (Placebo Comparator): 22 g/day placebo powder for 12 weeks
  Interventions: Dietary Supplement: Placebo Powder

INTERVENTIONS:
Dietary Supplement: Blueberry Powder — 22 g/day freeze-dried blueberry powder for 12 weeks
  Arms: Blueberry
Dietary Supplement: Placebo Powder — 22 g/day placebo powder for 12 weeks
  Arms: Control

SUMMARY:
Postmenopausal women are at an increased risk of developing cardiovascular disease (CVD) largely due to accelerated aging-related modifications to vascular health following menopause. The vascular endothelium is responsible for producing chemicals that are essential for proper vasodilation and blood flow and therefore is involved in maintaining normal blood pressure. A major modification that occurs during aging and is accelerated during menopause is termed vascular endothelial dysfunction which is characterized by impaired endothelium-dependent dilation. This can lead to increased blood pressure, atherosclerosis, and increased risk of CVD and death. Nitric oxide (NO) is a chemical produced by the endothelium and is essential for normal endothelial function and cardiovascular health. Vascular endothelial dysfunction is primarily caused by reduced NO bioavailability secondary to excessive oxidative stress. Approximately 3/4 of postmenopausal women have elevated blood pressure or hypertension which further worsens endothelial function and increases CVD risk through increased oxidative stress and inflammation. Blueberries are rich in phytochemicals including anthocyanins, phenolic acids, and pterostilbene. These phytochemicals and their metabolites are known to attenuate oxidative stress and inflammation. The overall goal of the current study is to assess the efficacy of blueberries to improve vascular endothelial dysfunction in this high-risk population and to gain insight into underlying mechanisms. 58 postmenopausal women with elevated blood pressure and stage 1-HTN will be asked to consume 22 grams freeze-dried blueberry powder or placebo powder per day for 12 weeks. Vascular endothelial function will be assessed at baseline and 12 weeks. Measurements indicative of vascular nitric oxide production, oxidative stress, inflammation, cardiometabolic health, cognitive function, and blueberry phytochemical metabolism will be measured at baseline and 12 weeks. Blood pressure will be assessed at baseline and 4, 8, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45-65 years
* Postmenopausal women (≥ 1 years postmenopausal; natural or surgical menopause; confirmed by measurement of estradiol at a level < 30 pg/mL and follicle-stimulating hormone at a level ≥ 30 mIU/mL)
* Elevated or stage 1-HTN (confirmed as resting seated systolic blood pressure < 120 or ≥ 139 mmHg and/or a diastolic blood pressure ≥ 90 mmHg using an average of 3 measurements, on 2 separate occasions - screening and baseline visits)
* Ability to provide informed consent

Exclusion Criteria:

* Systolic blood pressure < 120 or ≥ 139 mm Hg and/or diastolic blood pressure ≥ 90 mmHg
* Taking > 1 antihypertensive medication and/or taking the antihypertensive medication for < 3 months
* Diagnosed cancer, cardiovascular disease, diabetes, or gastrointestinal, kidney, liver, and/or pancreatic disease
* Triglycerides > 350 mg/dL, low-density lipoprotein cholesterol (LDL-C) ≥ 190 mg/dL, and/or taking a lipid-lowering medication
* Hormone replacement therapy use 6 months prior to study start
* Taking phosphodiesterase-5 inhibitors
* Weight change ≥ 3 kg in the past 3 months, actively trying to lose weight, or unwilling to remain weight stable throughout the study
* Current smokers or history of smoking in the past 12 months
* Binge and/or heavy drinker (>3 drinks on any given occasion and/or >7 drinks/week for women, and >4 drinks on any given occasion and/or >14 drinks/week for men)
* Body mass index < 18.5 or > 40 kg/m2
* Active infection or antibiotic therapy
* Allergies or contraindication to study treatments, pharmacological agents, or procedures

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 43 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent dilation | Baseline to 12 Weeks
  Assessed as brachial artery flow-mediated dilation in a study subset of participants
Blood pressure | Baseline to 12 weeks
  Assessed using an automated blood pressure monitor (SphgmoCor)

SECONDARY OUTCOMES:
Vascular oxidative stress | Baseline and 12 weeks
  Change in brachial artery flow-mediated dilation following acute infusion of ascorbic acid (a dose known to scavenge superoxide) as an index of vascular oxidative stress in a study subset of participants
Endothelial cell nitric oxide production, oxidative stress, and inflammation | Baseline and 12 weeks
  Protein expression markers will be measured by quantitative immunofluorescence in biopsied venous endothelial cells in a study subset of participants
Systemic markers of cardiometabolic health | Baseline and 12 weeks
  Circulating markers of lipid and glucose metabolism, nitric oxide, and inflammation
Plasma blueberry polyphenol metabolites | Baseline and 12 weeks
  Targeted analysis of plasma metabolites by GC-MS and LC-MS
Endothelium-independent dilation | Baseline to 12 weeks
  Assessed as brachial artery diameter responses to sublingual nitroglycerin in a study subset of participants
Augmentation index | Baseline to 12 weeks
  Arterial stiffness assessed as augmentation index using the SphygmoCor XCEL
Pulse wave velocity | Baseline to 12 weeks
  Arterial stiffness assessed as carotid-femoral pulse wave velocity using the SphygmoCor XCEL
Gut microbiota | Baseline to 12 weeks
  Determine the effects on stool sample microbial populations

OTHER OUTCOMES:
Processing speed | Baseline and 12 weeks
  Exploratory measures assessed using the NIH Cognitive Toolbox iPad app
Language | Baseline and 12 weeks
  Exploratory measures assessed using the NIH Cognitive Toolbox iPad app
Working memory | Baseline and 12 weeks
  Exploratory measures assessed using the NIH Cognitive Toolbox iPad app
Executive function and attention | Baseline and 12 weeks
  Exploratory measures assessed using the NIH Cognitive Toolbox iPad app
Episodic memory | Baseline and 12 weeks
  Exploratory measures assessed using the NIH Cognitive Toolbox iPad app
Peripheral blood mononuclear cell inflammation and oxidative stress | Baseline and 12 weeks
  Exploratory measures analyzed by gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A. Johnson, PhD, RDN, Principal Investigator — Department of Food Science and Human Nutrition, Colorado State University
Locations (1):
- Department of Food Science and Human Nutrition, Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson SA, Figueroa A, Navaei N, Wong A, Kalfon R, Ormsbee LT, Feresin RG, Elam ML, Hooshmand S, Payton ME, Arjmandi BH. Daily blueberry consumption improves blood pressure and arterial stiffness in postmenopausal women with pre- and stage 1-hypertension: a randomized, double-blind, placebo-controlled clinical trial. J Acad Nutr Diet. 2015 Mar;115(3):369-377. doi: 10.1016/j.jand.2014.11.001. Epub 2015 Jan 8. PMID 25578927
- [Derived] Woolf EK, Terwoord JD, Litwin NS, Vazquez AR, Lee SY, Ghanem N, Michell KA, Smith BT, Grabos LE, Ketelhut NB, Bachman NP, Smith ME, Le Sayec M, Rao S, Gentile CL, Weir TL, Rodriguez-Mateos A, Seals DR, Dinenno FA, Johnson SA. Daily blueberry consumption for 12 weeks improves endothelial function in postmenopausal women with above-normal blood pressure through reductions in oxidative stress: a randomized controlled trial. Food Funct. 2023 Mar 20;14(6):2621-2641. doi: 10.1039/d3fo00157a. PMID 36847333
- See also: Related Info — http://www.fshn.chhs.colostate.edu/research/FFHH/index.aspx